CLINICAL TRIAL: NCT04792944
Title: Cerebral Aneurysms: a Retrospective Study on the Experience in Our Hospital With a Comparative Analysis Between the Different Techniques Used in Its Treatment
Brief Title: Brain Aneurysms: Utility of Cisternal Urokinase Irrigation
Acronym: BA&UK
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: CEIm 17-07-2019
Record Dates: First submitted 2021-03-07; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Vasospasm, Cerebral; Hydrocephalus
Keywords: Aneurysm; Subarachnoid haemorrhage; Fibrinolytic Therapy; Intracisternal fibrinolysis; Cerebral vasospasm; Delayed ischemic neurological deficit
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Hydrocephalus; Aneurysm | interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- No treatment: Those are the patients that do not receive any treatment for the aneurysm, neither endovascular nor surgical
- External ventricular drain only with neither embolization nor clipping: These patients will be treated with an external ventricular drain only with neither embolization nor clipping
  Interventions: Procedure: External ventricular drain
- Embolization: These patients will be treated endovascularly
  Interventions: Procedure: Endovascular treatment
- Programmed surgical clipping: These patients will be treated no on an emergency basis with surgical clipping of an aneurysm that has bled
  Interventions: Procedure: Clipping
- Emergency surgical clipping with cisternal urokinase administration: These patients with undergo emergency surgical clipping with cisternal urokinase administration
  Interventions: Drug: Urokinase; Procedure: Clipping
- Patients with incidental brain aneurysm discovery with no SAH and programmed aneurysm clipping: This group will include patients with incidental brain aneurysm discovery with no SAH and programmed aneurysm clipping
  Interventions: Procedure: Clipping

INTERVENTIONS:
Drug: Urokinase — Washing the subarachnoid clot induced by a subarachnoid haemorrhage aneurysmal bleeding with urokinase after aneurysm clipping
  Other Names: Aneurysm clipping plus cisternal lavage with Urokinase
  Groups: Emergency surgical clipping with cisternal urokinase administration
Procedure: Endovascular treatment — Aneurysm treatment through endovascular methods
  Groups: Embolization
Procedure: Clipping — Surgical clipping of brain aneurysms
  Groups: Emergency surgical clipping with cisternal urokinase administration; Patients with incidental brain aneurysm discovery with no SAH and programmed aneurysm clipping; Programmed surgical clipping
Procedure: External ventricular drain — Insertion of an external ventricular drain to treat acute hydrocephalus
  Groups: External ventricular drain only with neither embolization nor clipping

SUMMARY:
Despite the efforts made in its treatment, aneurysmal subarachnoid haemorrhage continues to induce high mortality and morbidity rates. Today there are treatment protocols in all hospitals. The vast majority prefer, whenever possible, the endovascular route, given its lesser aggressiveness and morbidity.

Although embolization prevents aneurysm' rebleeding, it does remove the subarachnoid blood clot. Therefore, it does not modify the evolution, incidence and severity of vasospasm.

The idea is to carry out a 10-year retrospective study classifying patients into five groups based on the type of treatment received, analyzing the results' differences. The aim is to improve what is done as much as possible and to be able to propose potential areas for improvement. Besides, this study will be the basis of a future prospective study, prepared without the current one's biases and errors.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage continues to have very high morbidity and mortality rates, despite the years elapsed and repeated attempts to reduce it.

Stabilizing the aneurysm by embolization or surgical clipping leaves unresolved the vasospasm, responsible for ischemic brain damage, causing neurological sequelae and cognitive impairment.

It has long been known that the deoxyhemoglobin liberated from the extravasated red blood cells retained in the subarachnoid clot is the leading cause of vasospasm. Different routes have been tried to minimize its deleterious effects, such as copious lavage of the skull base cisterns, lysing the subarachnoid clot with urokinase or rtPA, administration of vitamin C, iron chelators, or superoxydodismutase-like drugs.

The volume of subarachnoid hemorrhage was soon correlated with the vasospasm severity. Once this fact was known in the 1980s and 1990s, cisternal lavage was used extensively during aneurysms' surgical clipping. Clots located in the subarachnoid space were lysed with urokinase or rtPA (recombinant tissue plasminogen activator), showing positive effects, particularly evident for the most severe bleeds, those with Fisher's grades of 3 or higher.

However, the introduction of embolization changed the treatment paradigm. As the craniotomy is not carried out, the cisterns are not usually washed, which controls the rebleeding but not the vasospasm. To date, we are not aware of any study that compares the effect on vasospasm of embolization versus clipping of aneurysms with lavage of the cisterns using thrombolytic agents.

In the Neurosurgery Department of our Hospital, two periods can be identified in which the treatment of brain aneurysms has been carried out differently. In the first period between 2007 and 2011, the aneurysms were primarily subjected to embolization, and only if there was no indication for endovascular treatment, surgical clipping was performed. In the second period, between 2012 and 2018, they were operated on an emergency basis with clip application and the skull base cisterns washed with urokinase. Embolization was considered if the surgical clipping was judged too risky.

The aim is to analyze these two periods and compare the mortality, morbidity, and vasospasm rates, the need for a cerebrospinal fluid diversion (temporary and definitive), and the final neurological and cognitive status for the different therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* harbour one or more saccular brain aneurysms
* with or without subarachnoid hemorrhage (SAH)
* multiple aneurysms

Exclusion Criteria:

* absence of brain fusiform, traumatic or mycotic aneurysms
* SAH due to other causes (trauma, anticoagulation, antiplatelet medication, arteriovenous malformation, or tumor)
* any medical, neurological, or psychiatric condition that would impair patient's evaluation
* past medical history of bleeding disorders or liver diseases altering the coagulation
* anticoagulation
* platelet count <10x109/L
* prothrombin time >15 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study of all brain aneurysms treated in our Hospital since 2007
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Vasospasm | 21 days
  Presence and severity of vasospasm
Cerebrospinal fluid diversion | 1 year
  Need for temporary or definitive cerebrospinal fluid diversion
Mortality rate | 1 year
  Mortality rate in each group of patients
Outcome | 1 year
  Glasgow Outcome Score (GOSE) at discharge, 6 and 12 months posttreatment

SECONDARY OUTCOMES:
Aneurysm regrowth | 10 years
  Aneurysm regrowth on follow-up after each tipe of treatment
Aneurysm rebleed | 10 years
  Aneurysm rebleed on follow-up after each tipe of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Teresa V Moratal, Nurse, Study Chair — Hospital General Universitario Valencia
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Mufti F, Amuluru K, Damodara N, El-Ghanem M, Nuoman R, Kamal N, Al-Marsoummi S, Morris NA, Dangayach NS, Mayer SA. Novel management strategies for medically-refractory vasospasm following aneurysmal subarachnoid hemorrhage. J Neurol Sci. 2018 Jul 15;390:44-51. doi: 10.1016/j.jns.2018.02.039. Epub 2018 Feb 23. PMID 29801906
- [Result] Arakawa Y, Kikuta K, Hojo M, Goto Y, Yamagata S, Nozaki K, Hashimoto N. Milrinone reduces cerebral vasospasm after subarachnoid hemorrhage of WFNS grade IV or V. Neurol Med Chir (Tokyo). 2004 Aug;44(8):393-400; discussion 401. doi: 10.2176/nmc.44.393. PMID 15508346
- [Result] Arthur AS, Fergus AH, Lanzino G, Mathys J, Kassell NF, Lee KS. Systemic administration of the iron chelator deferiprone attenuates subarachnoid hemorrhage-induced cerebral vasospasm in the rabbit. Neurosurgery. 1997 Dec;41(6):1385-91; discussion 1391-2. doi: 10.1097/00006123-199712000-00028. PMID 9402590
- [Result] Asano T. Oxyhemoglobin as the principal cause of cerebral vasospasm: a holistic view of its actions. Crit Rev Neurosurg. 1999 Sep 24;9(5):303-318. doi: 10.1007/s003290050147. PMID 10525849
- [Result] Ayer RE, Zhang JH. Oxidative stress in subarachnoid haemorrhage: significance in acute brain injury and vasospasm. Acta Neurochir Suppl. 2008;104:33-41. doi: 10.1007/978-3-211-75718-5_7. PMID 18456995
- [Result] Barbosa MD, Arthur AS, Louis RH, MacDonald T, Polin RS, Gazak C, Kassell NF. The novel 5-lipoxygenase inhibitor ABT-761 attenuates cerebral vasospasm in a rabbit model of subarachnoid hemorrhage. Neurosurgery. 2001 Nov;49(5):1205-12; discussion 1212-3. doi: 10.1097/00006123-200111000-00032. PMID 11846914
- [Result] Bilginer B, Onal MB, Narin F, Soylemezoglu F, Ziyal IM, Ozgen T. The effects of intravenous cilostazol and nimodipine on cerebral vasospasm after subarachnoid hemorrhage in an experimental rabbit model. Turk Neurosurg. 2009 Oct;19(4):374-9. PMID 19847758
- [Result] Dalbayrak S, Altas M, Arslan R. The effects of timing of aneurysm surgery on vasospasm and mortality in patients with subarachnoid hemorrhage. Acta Neurol Belg. 2011 Dec;111(4):317-20. PMID 22368972
- [Result] Ding X, Wang ZG, Wang CW, Wang YH. [Timing of treatment on the prognosis of poor-grade aneurysmal subarachnoid hemorrhage patients]. Zhonghua Yi Xue Za Zhi. 2012 Dec 4;92(45):3211-4. Chinese. PMID 23328469
- [Result] Dorhout Mees SM, Molyneux AJ, Kerr RS, Algra A, Rinkel GJ. Timing of aneurysm treatment after subarachnoid hemorrhage: relationship with delayed cerebral ischemia and poor outcome. Stroke. 2012 Aug;43(8):2126-9. doi: 10.1161/STROKEAHA.111.639690. Epub 2012 Jun 14. PMID 22700527
- [Result] Findlay JM. A randomized trial of intraoperative, intracisternal tissue plasminogen activator for the prevention of vasospasm. Neurosurgery. 1995 Nov;37(5):1026-7. doi: 10.1227/00006123-199511000-00031. No abstract available. PMID 8559330
- [Result] Gorski R, Zabek M, Jarmuzek P. Influence of intraoperative using of recombinant tissue plasminogen activator on the development of cerebral angiospasm after subarachnoid haemorrhage in patients with ruptured intracranial aneurysms. Neurol Neurochir Pol. 2000;34(6 Suppl):41-7. PMID 11452854
- [Result] Hamada J, Mizuno T, Kai Y, Morioka M, Ushio Y. Microcatheter intrathecal urokinase infusion into cisterna magna for prevention of cerebral vasospasm: preliminary report. Stroke. 2000 Sep;31(9):2141-8. doi: 10.1161/01.str.31.9.2141. PMID 10978043
- [Result] Handa Y, Kaneko M, Takeuchi H, Tsuchida A, Kobayashi H, Kubota T. Effect of an antioxidant, ebselen, on development of chronic cerebral vasospasm after subarachnoid hemorrhage in primates. Surg Neurol. 2000 Apr;53(4):323-9. doi: 10.1016/s0090-3019(00)00168-3. PMID 10825515
- [Result] Hanggi D, Steiger HJ. The influence of cisternal and ventricular lavage on cerebral vasospasm in patients suffering from subarachnoid hemorrhage: analysis of effectiveness. Acta Neurochir Suppl. 2011;110(Pt 2):95-8. doi: 10.1007/978-3-7091-0356-2_17. PMID 21125452
- [Result] Hirashima Y, Endo S, Horie Y, Kurimoto M. Indications for cisternal irrigation with urokinase in postoperative patients with aneurysmal subarachnoid haemorrhage. Br J Neurosurg. 1996 Oct;10(5):477-81. doi: 10.1080/02688699647113. PMID 8922707
- [Result] Hosoda K, Fujita S, Kawaguchi T, Shose Y, Hamano S, Iwakura M. Effect of clot removal and surgical manipulation on regional cerebral blood flow and delayed vasospasm in early aneurysm surgery for subarachnoid hemorrhage. Surg Neurol. 1999 Jan;51(1):81-8. doi: 10.1016/s0090-3019(97)00508-9. PMID 9952128
- [Result] Inagawa T, Yamamoto M, Kamiya K. Effect of clot removal on cerebral vasospasm. J Neurosurg. 1990 Feb;72(2):224-30. doi: 10.3171/jns.1990.72.2.0224. PMID 2295920
- [Result] Jito J, Nakasu Y, Nakasu S, Hatsuda N, Matsuda M. Tissue plasminogen activator levels after single intracisternal injection in patients with subarachnoid hemorrhage. Neurol Med Chir (Tokyo). 2004 Feb;44(2):55-60; discussion 60. doi: 10.2176/nmc.44.55. PMID 15018324
- [Result] Kajimoto Y, Ohta T, Kuroiwa T. Comparison of intrathecally administered urokinase, tissue-type plasminogen activator, and combination of urokinase and lysine-plasminogen for clot lysis after experimental subarachnoid hemorrhage in dogs. Neurosurgery. 1997 Mar;40(3):572-7. doi: 10.1097/00006123-199703000-00029. PMID 9055298
- [Result] Kawakami M, Kodama N, Toda N. Suppression of the cerebral vasospastic actions of oxyhemoglobin by ascorbic acid. Neurosurgery. 1991 Jan;28(1):33-9; discussion 39-40. doi: 10.1097/00006123-199101000-00006. PMID 1704491
- [Result] Kodama N, Matsumoto M, Sasaki T, Konno Y, Sato T. Cisternal irrigation therapy with urokinase and ascorbic acid for prevention of vasospasm. Acta Neurochir Suppl. 2001;77:171-4. doi: 10.1007/978-3-7091-6232-3_36. No abstract available. PMID 11563280
- [Result] Li YH, Guo K, Zi XH, Song Z. [Combining exchange of cerebrospinal fluid with small dose of urokinase injection for subarachnoid hemorrhage]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2005 Apr;30(2):217-20. Chinese. PMID 15898439
- [Result] Macdonald RL, Weir BK. A review of hemoglobin and the pathogenesis of cerebral vasospasm. Stroke. 1991 Aug;22(8):971-82. doi: 10.1161/01.str.22.8.971. PMID 1866764
- [Derived] De BP, Rosenberg JB, Selvan N, Wilson I, Yusufzai N, Greco A, Kaminsky SM, Heier LA, Ricart Arbona RJ, Miranda IC, Monette S, Nair A, Khanna R, Crystal RG, Sondhi D. Assessment of Safety and Biodistribution of AAVrh.10hCLN2 Following Intracisternal Administration in Nonhuman Primates for the Treatment of CLN2 Batten Disease. Hum Gene Ther. 2023 Sep;34(17-18):905-916. doi: 10.1089/hum.2023.067. PMID 37624739